CLINICAL TRIAL: NCT00210171
Title: Multicentric Phase II Study of Concomitant Chemo-radiotherapy in Locally Advanced Non Small Cell Lung Cancer, With :- Induction Chemotherapy by Cisplatin - Docetaxel- Concomitant Chemo-radiotherapy by Weekly Cisplatin - Docetaxel- Consolidation Chemotherapy by Docetaxel
Brief Title: Concomitant Chemo-radiotherapy in Locally Advanced Non Small Cell Lung Cancer
Acronym: BIB 01
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was withdrawn due to logistic issues.
Sponsor: Institut Bergonié (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Purpose: Treatment
Other Study IDs: IB2004-20; BIB-01
Record Dates: First submitted 2005-09-12; First posted 2005-09-21 (Estimated); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Carcinoma; Stage IIIA Non Small Cell Lung; Stage IIIB Non-Small-Cell Lung; Concomitant chemo-radiotherapy; Consolidation chemotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Toxicity : Time to progression, 1 and 2 years survival

SUMMARY:
Feasibility of pragmatic concomitant chemo-radiotherapy association with 1 cycle of Induction chemotherapy, weekly chemo-radiotherapy, and consolidation chemotherapy.

ELIGIBILITY:
Inclusion criteria:

Histologically or cytologically confirmed newly diagnosed, untreated, unresectable stage IIIA or stage IIIB non-small cell lung cancer Not scheduled for curative cancer surgery No pleural effusion At least 1 bidimensionally or unidimensionally measurable lesion Age 18 years et 70 years; Performance Status < 2 Loss of weight < 10 % in past 6 months life expectancy 12 weeks; Bilirubin normal ASAT (SGOT) et ALAT (SGPT) 1,5 times upper limit of normal; Alcalin phosphatases 5 times upper limit of normal; Créatinin 1,5 x times upper limit of normal; Absolute neutrophil count greater than 2.109/l; Platelet count greater than 100.109/l; Hémoglobin ³ 10 g/ dl; Respiratory function : FEV1>50% write Consent

Exclusion criteria:

Pregnant or nursing; Fertile patients who don't used effective contraception; No other malignancy within past 5 years except inactive carcinoma in situ of the cervix or nonmelanoma skin cancer ; Neuropathy grade NCI-CTC 2; Past thoracic radiotherapy; Past chemotherapy, immunotherapy or biologic therapy for non small cell lung cancer ; Respiratory deficiency FEV1 < 45% ; Hypersensibility to docetaxel or cisplatin; At least 4 weeks since other concurrent investigational agents;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2004-05 (Actual); Primary Completion 2004-05 (Actual); Study Completion 2004-05 (Actual)

PRIMARY OUTCOMES:
Objective response | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: François CHOMY, MD, Principal Investigator — Institut Bergonié
Locations (7):
- France (7):
  - Centre de radiothérapie d'Agen, Agen
  - Clinique Tivoli, Bordeaux
  - Polyclinique Bordeaux Nord, Bordeaux
  - Centre Hospitalier Universitaire de Bordeaux, Bordeaux
  - Institut Bergonié - Centre Régional de Luttre Contre le Cancer de Bordeaux et du Sud Ouest, Bordeaux
  - Hôpital Robert Boulin, Libourne
  - Clinique Francheville, Périgueux

IPD SHARING:
Plan to Share IPD: No